CLINICAL TRIAL: NCT03616171
Title: A Sleep Intervention (SLEEP-Extend) for Young Adults At-Risk for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ashley Coombe, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00105390; 5P30DK111024-02 (NIH)
Record Dates: First submitted 2018-07-23; First posted 2018-08-06 (Actual); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Sleep Behavior; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Prospective, randomized and unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Intervention Group (SLEEP-Extend intervention): The SLEEP-Extend intervention consists of two components:
  1. One education session (5-10 minutes) consisting of strategies for sleep hygiene which is the routine for going to sleep (an investigator-developed brochure and information based on recommendations from the American Academy of Sleep Medicine and the National Sleep Foundation will be given and reviewed with the subject)
  2. Instructions on extending time in bed by at least one hour but can be up to 2 hours total per night for 4 weeks which can be accomplished by either going to bed earlier or staying in bed later (subject will decide what works best for them).
  Interventions: Behavioral: SLEEP-Extend intervention
- Control Group (Other): Control group: consists of One educational session (5-10 minutes) consisting of safety practices used for an urban environment (a safety brochure and safety information will be given and reviewed with the subject)
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: SLEEP-Extend intervention — 1. One education session (5-10 minutes) consisting of strategies for sleep hygiene which is the routine for going to sleep
  2. Instructions on extending time in bed by at least one hour but can be up to 2 hours total per night for 4 weeks which can be accomplished by either going to bed earlier or staying in bed later
  Arms: Interventional Group
Other: Control — Control group will receive 1. One educational session (5-10 minutes) consisting of safety practices used for an urban environment (a safety brochure and safety information will be given and reviewed with the subject)
  Arms: Control Group

SUMMARY:
The study is a prospective unblinded randomized trial to evaluate the feasibility of conducting a sleep extension intervention trial and the sleep extension intervention among the young adults. The study also wants to assess whether a sleep-extension intervention has an impact on the insulin resistance levels of young adults. The intervention consists of an education session and to extend the sleep time at least one hour but can be up to 2 hours per night for 4 weeks.

DETAILED DESCRIPTION:
Insulin Resistance has been shown to put a person at risk for developing Type II diabetes. There is a correlation between sleep deprivation and insulin resistance.The study wants to assess the feasibility by enrolling 20 subjects in a year. The study also wants to assess the feasibility of the sleep extension intervention among young adults by examining the number of subjects that are randomized to intervention arm will complete the study.

Another intent of the study is to examine how sleep behaviors affect risks for developing type 2 diabetes and to determine their willingness to participate in a 4-week home-based program (intervention) focused on personal sleep behaviors.

Subjects enrolled in the study and are randomized to intervention group and control group. The intervention group will receive one education session consisting of strategies for sleep hygiene which is the routine for going to sleep and instructions on extending time in bed by at least one hour but can be up to 2 hours total per night for 4 weeks. At the end of 4 weeks subjects will have a blood draw and will complete the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age must be 18-25 years old
* Self-report short sleep
* BMI ≥ 30 (the World Health Organization's classification of being obese)
* Insulin Resistance determined by serum analysis
* Be willing to extend time in bed by one hour total per night
* Read and speak English.

Exclusion Criteria:

* Night shift worker;
* Sleep disorder diagnosis;
* Medical diagnosis of diabetes or pre-diabetes;
* Currently pregnant or lactating or with history of gestational diabetes;
* Actively participating in a weight loss program;
* Hospitalization in past 3 months for any medical or psychiatric condition;
* Having a major chronic illness (e.g. cancer, Lupus)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Coombe, PhD, RN, CNE, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Georgia State University, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between August 30, 2017 and April 2, 2018 from Georgia State University in Atlanta, Georgia.
Pre-assignment Details: A total of 19 individuals consented to take part in the study, of which 13 did not meet eligibility criteria during the screening process, resulting in 6 participants who were randomized to a study arm.
Groups:
- SLEEP-Extend Intervention: Participants receiving one educational session consisting of strategies for sleep hygiene and instruction to increase time in bed by a total of one hour.
- Control Group: Participants receiving one educational session consisting of safety practices used for an urban environment.
Period: Overall Study
Arm/Group | SLEEP-Extend Intervention | Control Group
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SLEEP-Extend Intervention | Control Group | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (0.82) | 21.5 (4.95) | 19.83 (2.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 0 | 3
  White | 1 | 1 | 2
  Persian | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 2 | 6
Marital Status [Count of Participants; unit: Participants]
  Single | 4 | 2 | 6
  Married | 0 | 0 | 0
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Enrollments in the Study Over One Year
Description: Feasibility of the study is assessed by number of enrollments in the study over a one year period. Study proposes to enroll minimum 20 subjects to meet the feasibility of the study.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | SLEEP-Extend Intervention | Control Group
Number analyzed (Participants) | 4 | 2
Participants | 4 | 2

2. Primary Outcome: Number of Participants Enrolled in the Intervention Arm Who Complete the Study
Description: Feasibility of the SLEEP-Extend intervention among young adults is measured by number of participants enrolled in the intervention arm that received the intervention and completed the study required protocols for the study duration of 4 weeks.
Time Frame: Week 4
Population: Only participants in the intervention arm are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | SLEEP-Extend Intervention
Number analyzed (Participants) | 4
Participants | 4

3. Secondary Outcome: Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) Scores
Description: The HOMA-IR score is used to measure severity of insulin resistance, though normal insulin resistance varies depending on the population. HOMA-IR is calculated as blood glucose level (nmol/L) multiplied by insulin level (microU/L), divided by 22.5. Elevated values indicate insulin resistance. A cutoff score of HOMA-IR < 2.1 is considered normal and HOMA-IR ≥ 2.1 is considered to be evidence of insulin resistance.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | SLEEP-Extend Intervention | Control Group
Number analyzed (Participants) | 4 | 2
HOMA-IR score
  Baseline | 5.73 (3.81) | 4.33 (0.94)
  Week 4 | 6.55 (5.47) | 5.13 (1.54)

4. Secondary Outcome: Hours of Sleep
Description: Using wrist actigraphy, this study will objectively monitor each participant's 24-hour sleep-wake cycle to obtain average sleep duration (total sleep time) over one week.
Time Frame: Over a 1 week period at Baseline, and over a 1 week period at Week 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SLEEP-Extend Intervention | Control Group
Number analyzed (Participants) | 4 | 2
hours
  Baseline | 5.18 (0.55) | 5.78 (0.01)
  Week 4 | 5.63 (0.92) | 6.72 (0.41)

5. Secondary Outcome: Number of Participants Extending Sleep
Description: Sleep extension is assessed as the number of participants extending their nightly sleep by 1 to 2 hours from the baseline visit to the week 4 visit, as monitored using wrist actigraphy to measure each participant's 24-hour sleep-wake cycle to obtain average sleep duration (total sleep time) over one week.
Time Frame: Over a 1 week period at Baseline, and over a 1 week period at Week 4
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Participants receiving one educational session consisting of safety practices for an urban environment.
Arm/Group | SLEEP-Extend Intervention | Control Group
Number analyzed (Participants) | 4 | 2
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time of consenting to take part in the study throughout the 4 week study duration.
Arm/Group | SLEEP-Extend Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-04-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03616171/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT03616171/Prot_SAP_001.pdf